CLINICAL TRIAL: NCT05633823
Title: The Effect of Mobile Application Game Training Designed for Children With Asthma on Asthma Management
Brief Title: The Effect of Mobile Application Game Training Designed for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Ass. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022/13
Record Dates: First submitted 2022-11-18; First posted 2022-12-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-04

CONDITIONS: Asthma in Children; Life Style; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game group (Experimental): Children and parents will be introduced to mobile application game training and they will be provided to download the application to their mobile device or tablet. The data collection forms will be applied again immediately after the children complete each part of the game, 4 months and 6 months after the training.
  Interventions: Other: Mobile Application Game Training
- Control group (No Intervention): No application will be made to children and parents, and the forms will be re-applied 4 months and 6 months after the first application of the data collection forms.

INTERVENTIONS:
Other: Mobile Application Game Training — Mobile application game training can be used interactively with smartphones and tablets.
  * A user account will be created after the application is downloaded to the mobile phone/tablet.
  * After logging into the application, the map of the game will be displayed.
  * The game will start with the first level of the game consisting of 5 levels.
  * At each level, first of all, educational videos prepared in the form of short (1-2 minutes) animations will be watched. The number of videos varies between 1 and 3.
  * After watching the videos, interactive games will be played.
  * Children are required to complete each stage in the game, and each stage is planned to take approximately 7-10 minutes.
  * After passing the first level, children will be able to move on to the next level of games and will not be able to move on to the next level until the previous level is finished.
  Arms: Game group

SUMMARY:
The aim of this research is to examine the effect of mobile application game training designed for children aged 8-16 years on asthma management and quality of life. The population of the study will be children in the 8-12 age group who applied to the Mersin Pediatric Allergy, Asthma and Immunology Specialist's clinic, and the sample will consist of 78 children with asthma who meet the criteria for inclusion in the research. This age group has problems in solving abstract problems, it is necessary to embody it in order to facilitate the understanding of the disease process. Therefore, it is important to embody the training given in the increase of self-management related to the disease process of this age group. While determining the sample size of the study, Arıkan-Ayyıldız et al. (2016) based on the scientific study named "Efficacy of asthma education program on asthma control in children with uncontrolled asthma". In the Arıkan-Ayyıldız study, it was reported that the total mean score of "ACT" (Asthma Control Test-Asthma Control Test) was 13.8±3.4 in the experimental group and 15.6±3.2 in the control group. As a result of the Power analysis (G*Power 3.1.9.2) made according to these data; effect size = 0.78, with 95% confidence interval, 95% power, it was calculated that a total of 72 children with asthma, at least 36 in each group, should be included. Considering that there may be dropout and confounders during the research process, the number of groups was increased by 10%. The sample of the research; was a total of 78 children, including 39 children in each intervention group.

In collecting research data; the Child and Parent Information Form, Inhaler Usage Skills Evaluation Form, Asthma Symptom and Treatment Need Scoring, DISABKIDS Asthma Scale will be used. A statistical package program (SPSS 20) will be used in the analysis of the research data. The statistical significance level was determined as 0.05. Kolmogorov-Smirnov will be used in the normality analysis of dependent variables. Chi-square and mean-to-means comparison tests will be used to determine the similarity of the groups. Appropriate parametric or non-parametric tests will be used according to the distribution's normality in comparing the means between groups and within groups.

DETAILED DESCRIPTION:
* Data will be collected in the waiting room after the child is examined at the clinic. In data collection, the pediatric patients who applied to the clinic of the Pediatric Allergy, Asthma and Immunology Specialist who met the inclusion criteria of the study and agreed to participate in the study, and their parents, who were diagnosed with asthma at least one year ago, will be informed about the purpose of the study and their parents, and their verbal and written consent will be obtained.
* Randomization will be provided by randomly and evenly dividing the patients who meet the sample selection criteria into 2 groups (1st experimental group, 2nd group control group) through a computer program (http://www1.assumption.edu/users/avadum/applets/). RandAssign/GroupGen.html).
* The data collection forms in the research will be applied to the children and parents in the sample group.
* Mobile application game training will be introduced to the children and parents in the experimental group and they will be provided to download the application to their mobile device or tablet.
* Data collection forms will be re-applied immediately after children complete one round of the game, 4 months and 6 months after the training.
* No application will be made to the children and parents in the control group, and the forms will be re-applied 4 months and 6 months after the first application of the data collection forms.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 8-12
* Having been diagnosed with asthma according to ICD-10 in the last year
* Being on an inhaled corticosteroid or leukotriene antagonist (LTA)
* Not having any other chronic disease
* Having a phone/tablet with a parent or a mobile gameplay feature
* No communication, mental or neurological problems
* Volunteering to participate in the study
* Not being obese (3-90% percentile value)
* Moderate or severe asthma according to asthma severity classification

Exclusion Criteria:

* Not to be between the ages of 8-12
* Not having been diagnosed with asthma according to ICD-10 in the last year
* Having had a viral infection in the last two weeks
* Not using inhaled corticosteroids
* Having another chronic disease
* Not having a parent or a phone/tablet with mobile gameplay feature
* Having a communication, mental or neurological problem
* Not volunteering to participate in the study
* Being obese (more than 90% percentile)
* Mild asthma according to asthma severity classification

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Using Inhaler Skill Evaluation Form | 1 day
  The Skills Evaluation Form was prepared by using the brochure and literature prepared by the Turkish Respiratory Research Association Inhalation Therapies Working Group, based on correct inhalation techniques. The form consists of 10 skill steps in which the skills of using inhalation devices used in the treatment of asthma are evaluated. There are 4 subgroups in the form, including metered dose inhaler (MDI), turbohaler, discus and aerolizer type instruments. According to the scoring system used in the researches, "0" points are given for "Wrong" or skipped steps, and "1" points are given for "Correct" steps. A score between 0 and 10 is obtained by summing the scores obtained from all the steps evaluated by the direct observation method. The form will be filled by the same researcher using the observation method. In cases where more than one inhaler device is used, the average score will be taken. In the evaluation of the form; A high score indicates a good level of inhaler use.
Asthma Symptom and Need for Treatment Scoring | 1 day
  This form was created to monitor the changes in the clinical symptoms of children with asthma (Liu et al., 2007; Al Aloola et al., 2017). It will be given at the beginning of the study so that the child and their parents can record their asthma symptoms. in form; respiratory tract complaints and asthma symptoms (cough, wheezing, shortness of breath, frequent breathing, phlegm, night cough), nasal complaints/ rhinitis symptoms (runny nose, congestion, sneezing, itchy eyes, watery eyes and itchy nose) no symptoms according to the degree of complaint It is scored as 0 if it is light, 2 if it is moderate, and 3 if it is heavy. These symptom scores will be calculated as asthma symptom score (ASS) and rhinitis symptom score (RSS) by giving the mean value. Total symptom score (TSS) will be taken as the sum of ASS and RSS.
DISABKIDS Asthma Scale | 1 day
  The questions in the scale are evaluated using 1-5 point Likert type questions. "1" represents the most negative rating and "5" represents the most positive rating. The score weights of the questions are equal. The total score for all items is between 11-55. The scale has two sub-dimensions as effect and anxiety. There are 6 questions in the effect dimension and 5 questions in the anxiety dimension. In addition, there is an additional symptom section consisting of three questions for symptom control. This section is not included in the scoring, it provides an idea about the patient's asthma status. It is thought that the higher the score the patient gets from the scale, the better the quality of life. The cronbach alpha value of the scale is 0.86

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sönmez Düzkaya, Principal Investigator — Tarsus University; Gamze Bozkul, Principal Investigator — Tarsus University
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Aloola NA, Nissen L, Alewairdhi HA, Al Faryan N, Saini B. Parents' asthma information needs and preferences for school-based asthma support. J Asthma. 2017 Nov;54(9):946-956. doi: 10.1080/02770903.2017.1281296. Epub 2017 Jan 17. PMID 28095117
- [Background] Arikan-Ayyildiz Z, Isik S, Caglayan-Sozmen S, Anal O, Karaman O, Uzuner N. Efficacy of asthma education program on asthma control in children with uncontrolled asthma. Turk J Pediatr. 2016;58(4):383-388. doi: 10.24953/turkjped.2016.04.006. PMID 28276210
- [Background] Bruggers CS, Baranowski S, Beseris M, Leonard R, Long D, Schulte E, Shorter A, Stigner R, Mason CC, Bedrov A, Pascual I, Bulaj G. A Prototype Exercise-Empowerment Mobile Video Game for Children With Cancer, and Its Usability Assessment: Developing Digital Empowerment Interventions for Pediatric Diseases. Front Pediatr. 2018 Apr 9;6:69. doi: 10.3389/fped.2018.00069. eCollection 2018. PMID 29686977
- [Background] Castro-Rodriguez JA, Forno E, Rodriguez-Martinez CE, Celedon JC. Risk and Protective Factors for Childhood Asthma: What Is the Evidence? J Allergy Clin Immunol Pract. 2016 Nov-Dec;4(6):1111-1122. doi: 10.1016/j.jaip.2016.05.003. Epub 2016 Jun 8. PMID 27286779
- [Background] Cheng J, Wang H, Zhang X, Guo H, Duan H. The factors of family management affecting asthma control status in school-age children with asthma in China. J Asthma. 2022 May;59(5):1041-1050. doi: 10.1080/02770903.2021.1895209. Epub 2021 Mar 22. PMID 33629923
- [Background] Cook KA, Modena BD, Simon RA. Improvement in Asthma Control Using a Minimally Burdensome and Proactive Smartphone Application. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):730-737.e1. doi: 10.1016/j.jaip.2016.03.005. Epub 2016 Apr 20. PMID 27107690
- [Background] Davis SR, Peters D, Calvo RA, Sawyer SM, Foster JM, Smith LD. A consumer designed smartphone app for young people with asthma: pilot of engagement and acceptability. J Asthma. 2021 Feb;58(2):253-261. doi: 10.1080/02770903.2019.1680997. Epub 2019 Nov 6. PMID 31691618
- [Background] Deniz PÖ, Abacıgil F, Uysal P. Çocuk ve Ergenlerde Disabkids Astım Modülünün Geçerlilik ve Güvenilirliği. 4. Uluslararası 22. Ulusal Halk Sağlığı Kongresi, 2020.
- [Background] Fedele DA, McConville A, Graham Thomas J, McQuaid EL, Janicke DM, Turner EM, Moon J, Abu-Hasan M. Applying Interactive Mobile health to Asthma Care in Teens (AIM2ACT): Development and design of a randomized controlled trial. Contemp Clin Trials. 2018 Jan;64:230-237. doi: 10.1016/j.cct.2017.09.007. Epub 2017 Oct 3. PMID 28986245
- [Background] Fedele DA, Thomas JG, McConville A, McQuaid EL, Voorhees S, Janicke DM, Abu-Hasan M, Chi X, Gurka MJ. Using Mobile Health to Improve Asthma Self-Management in Early Adolescence: A Pilot Randomized Controlled Trial. J Adolesc Health. 2021 Dec;69(6):1032-1040. doi: 10.1016/j.jadohealth.2021.06.011. Epub 2021 Jul 15. PMID 34274211
- [Background] Franzmair J, Diesner-Treiber SC, Voitl JJM, Voitl P. Effective German and English Language mHealth Apps for Self-management of Bronchial Asthma in Children and Adolescents: Comparison Study. JMIR Mhealth Uhealth. 2021 May 19;9(5):e24907. doi: 10.2196/24907. PMID 34009134
- [Background] Fuemmeler BF, Holzwarth E, Sheng Y, Do EK, Miller CA, Blatt J, Rosoff PM, Ostbye T. Mila Blooms: A Mobile Phone Application and Behavioral Intervention for Promoting Physical Activity and a Healthy Diet Among Adolescent Survivors of Childhood Cancer. Games Health J. 2020 Aug;9(4):279-289. doi: 10.1089/g4h.2019.0060. Epub 2020 May 8. PMID 32391734
- [Background] Gibson PG, Powell H, Coughlan J, Wilson AJ, Abramson M, Haywood P, Bauman A, Hensley MJ, Walters EH. Self-management education and regular practitioner review for adults with asthma. Cochrane Database Syst Rev. 2003;(1):CD001117. doi: 10.1002/14651858.CD001117. PMID 12535399
- [Background] Haktanir Abul M, Phipatanakul W. Severe asthma in children: Evaluation and management. Allergol Int. 2019 Apr;68(2):150-157. doi: 10.1016/j.alit.2018.11.007. Epub 2019 Jan 14. PMID 30648539
- [Background] Hsia B, Mowrey W, Keskin T, Wu S, Aita R, Kwak L, Ferastraoarou D, Rosenstreich D, Jariwala SP. Developing and pilot testing ASTHMAXcel, a mobile app for adults with asthma. J Asthma. 2021 Jun;58(6):834-847. doi: 10.1080/02770903.2020.1728770. Epub 2020 Feb 19. PMID 32046564
- [Background] Ivory, A.H., Ivory, J.D. (2017). On the Need for Developmental Perspectives in Research on the Potential Positive and Negative Health Effects of Digital Games. In: Marston, H., Freeman, S., Musselwhite, C. (eds) Mobile e-Health. Human-Computer Interaction Series. Springer
- [Background] Kelada L, Molloy CJ, Hibbert P, Wiles LK, Gardner C, Klineberg E, Braithwaite J, Jaffe A. Child and caregiver experiences and perceptions of asthma self-management. NPJ Prim Care Respir Med. 2021 Sep 9;31(1):42. doi: 10.1038/s41533-021-00253-9. PMID 34504105
- [Background] Kindi ZA, McCabe C, McCann M. Impact of Nurse-Led Asthma Intervention on Child Health Outcomes: A Scoping Review. J Sch Nurs. 2022 Feb;38(1):84-97. doi: 10.1177/10598405211003303. Epub 2021 Mar 24. PMID 33759614
- [Background] Kulikova A, Lopez J, Antony A, Khan DA, Persaud D, Tiro J, Ivleva EI, Nakamura A, Patel Z, Tipton S, Lloyd T, Allen K, Kaur S, Owitz MS, Pak RJ, Adragna MS, Chankalal R, Humayun Q, Lehman HK, Miller BD, Wood BL, Brown ES. Multivariate Association of Child Depression and Anxiety with Asthma Outcomes. J Allergy Clin Immunol Pract. 2021 Jun;9(6):2399-2405. doi: 10.1016/j.jaip.2021.02.043. Epub 2021 Mar 4. PMID 33677079
- [Background] Lin J, Wang W, Tang H, Huo J, Gu Y, Liu R, Chen P, Yuan Y, Yang X, Xu J, Sun D, Li N, Jiang S, Chen Y, Wang C, Yang L, Liu X, Yang D, Zhang W, Chen Z, Lin Q, Liu C, Zhou J, Zhou X, Hu C, Jiang P, Zhou W, Zhang J, Cai S, Qiu C, Huang M, Huang Y, Liu H; China Asthma Research Collaboration Network. Asthma Management Using the Mobile Asthma Evaluation and Management System in China. Allergy Asthma Immunol Res. 2022 Jan;14(1):85-98. doi: 10.4168/aair.2022.14.1.85. PMID 34983109
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Lv S, Ye X, Wang Z, Xia W, Qi Y, Wang W, Chen Y, Cai X, Qian X. A randomized controlled trial of a mobile application-assisted nurse-led model used to improve treatment outcomes in children with asthma. J Adv Nurs. 2019 Nov;75(11):3058-3067. doi: 10.1111/jan.14143. Epub 2019 Aug 12. PMID 31241192
- [Background] Lyons EJ, Baranowski T, Basen-Engquist KM, Lewis ZH, Swartz MC, Jennings K, Volpi E. Testing the effects of narrative and play on physical activity among breast cancer survivors using mobile apps: study protocol for a randomized controlled trial. BMC Cancer. 2016 Mar 9;16:202. doi: 10.1186/s12885-016-2244-y. PMID 26960972
- [Background] Masoli M, Fabian D, Holt S, Beasley R; Global Initiative for Asthma (GINA) Program. The global burden of asthma: executive summary of the GINA Dissemination Committee report. Allergy. 2004 May;59(5):469-78. doi: 10.1111/j.1398-9995.2004.00526.x. No abstract available. PMID 15080825
- [Background] Meyer R, Wang K, Yearley A, Grob S, Zeitlin J, Bloomfeld J, You M, Lee D, Bonner M, Shah N, Page K. Usability and Acceptability of the QuestLeukemia Mobile Application: A Pilot Study for An Educational and Psychological Intervention for Children with Chronic Illnesses. J Pediatr Hematol Oncol Nurs. 2022 May-Jun;39(3):137-142. doi: 10.1177/27527530221068422. Epub 2022 Jan 25. PMID 35467435
- [Background] Pearce N, Ait-Khaled N, Beasley R, Mallol J, Keil U, Mitchell E, Robertson C; ISAAC Phase Three Study Group. Worldwide trends in the prevalence of asthma symptoms: phase III of the International Study of Asthma and Allergies in Childhood (ISAAC). Thorax. 2007 Sep;62(9):758-66. doi: 10.1136/thx.2006.070169. Epub 2007 May 15. PMID 17504817
- [Background] Ramsey RR, Plevinsky JM, Kollin SR, Gibler RC, Guilbert TW, Hommel KA. Systematic Review of Digital Interventions for Pediatric Asthma Management. J Allergy Clin Immunol Pract. 2020 Apr;8(4):1284-1293. doi: 10.1016/j.jaip.2019.12.013. Epub 2019 Dec 21. PMID 31870809
- [Background] Real FJ, Beck AF, DeBlasio D, Zackoff M, Henize A, Xu Y, Davis D, Cruse B, Klein MD. Dose Matters: A Smartphone Application to Improve Asthma Control Among Patients at an Urban Pediatric Primary Care Clinic. Games Health J. 2019 Oct;8(5):357-365. doi: 10.1089/g4h.2019.0011. Epub 2019 Jun 3. PMID 31157983
- [Background] Sarasmita MA, Larasanty LPF, Kuo LN, Cheng KJ, Chen HY. A Computer-Based Interactive Narrative and a Serious Game for Children With Asthma: Development and Content Validity Analysis. J Med Internet Res. 2021 Sep 13;23(9):e28796. doi: 10.2196/28796. PMID 34515641
- [Background] Tark R, Metelitsa M, Akkermann K, Saks K, Mikkel S, Haljas K. Usability, Acceptability, Feasibility, and Effectiveness of a Gamified Mobile Health Intervention (Triumf) for Pediatric Patients: Qualitative Study. JMIR Serious Games. 2019 Sep 30;7(3):e13776. doi: 10.2196/13776. PMID 31573904
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Weinstein SM, Pugach O, Rosales G, Mosnaim GS, Orozco K, Pappalardo AA, Martin MA. Psychosocial Moderators and Outcomes of a Randomized Effectiveness Trial for Child Asthma. J Pediatr Psychol. 2021 Jul 20;46(6):673-687. doi: 10.1093/jpepsy/jsab011. PMID 33616185
- See also: Related Info — https://ginasthma.org/wp-content/uploads/2021/05/GINA-Main-Report-2021-V2-WMS.pdf
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/asthma